CLINICAL TRIAL: NCT02737033
Title: Effects of 800mg of Rhodiola Rosea in Attention in Adults With Attention-Deficit/Hyperactivity Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150426
Record Dates: First submitted 2016-03-07; First posted 2016-04-13 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Adults; Treatment; Rhodiola
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhodiola (Experimental): Rhodiola rosea 800mg single dose
  Interventions: Drug: Rhodiola
- Placebo (Placebo Comparator): placebo 800mg single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhodiola — Rhodiola rosea 800mg
  Other Names: Rhodiola rosea
  Arms: Rhodiola
Drug: Placebo — innocuous pill manufactured to mimic Rhodiola
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
This study evaluates the use of Rhodiola rosea in the attention of adults with Attention Deficit/Hyperactivity Disorder (ADHD). Half of participants will receive Rhodiola rosea 800mg, while the other half will receive 800mg of placebo.

DETAILED DESCRIPTION:
The evaluation of new therapies in adults with Attention Deficit/Hyperactivity Disorder (ADHD) may be clinically useful. Rhodiola rosea is an herbal medicine used for centuries in various medical conditions. Many randomized controlled trials have evaluated its usefulness in stress and fatigue. There were benefits in attention in some of these studies. Mild side effects and beneficial antioxidant properties make reasonable an assessment of its potential benefits in adults with ADHD. To our knowledge, Rhodiola rosea has never been studied in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5) diagnostic criteria for ADHD in Adults
* Intelligence Quotient (IQ) above 70
* Eligibility to Rhodiola rosea

Exclusion Criteria:

* clinical contraindication to Rhodiola rosea
* any unstable chronic illness without proper treatment (hypertension, heart, kidney or liver disease, etc)
* any significant neurological disease (delirium, dementia, epilepsy, AIDS, head trauma, multiple sclerosis, stroke, etc)
* unstable psychiatric comorbidities requiring immediate treatment (risk of suicide, current Substance Use Disorder, etc.)
* pregnant, nursing or absence of reliable contraception
* current use of nicotine (<30 days)
* use of anticoagulants
* current use of any psychoactive drug (<30 days)
* prior use of stimulants
* current or lifetime psychosis
* current or lifetime bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in Stop Signal Task | Baseline and 4 hours
  Change from baseline attention 4 hours after a single dose of Rhodiola 800mg or placebo

SECONDARY OUTCOMES:
Change in Wechsler Adult Intelligence Scale (WAIS) - Digit Span subtest | Baseline and 4 hours
  Change from baseline attention 4 hours after a single dose of Rhodiola 800mg or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Grevet, PhD, Principal Investigator — Hosptital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seixas M, Weiss M, Muller U. Systematic review of national and international guidelines on attention-deficit hyperactivity disorder. J Psychopharmacol. 2012 Jun;26(6):753-65. doi: 10.1177/0269881111412095. Epub 2011 Sep 24. PMID 21948938
- [Background] Meszaros A, Czobor P, Balint S, Komlosi S, Simon V, Bitter I. Pharmacotherapy of adult attention deficit hyperactivity disorder (ADHD): a meta-analysis. Int J Neuropsychopharmacol. 2009 Sep;12(8):1137-47. doi: 10.1017/S1461145709990198. Epub 2009 Jul 7. PMID 19580697
- [Background] Iovieno N, Dalton ED, Fava M, Mischoulon D. Second-tier natural antidepressants: review and critique. J Affect Disord. 2011 May;130(3):343-57. doi: 10.1016/j.jad.2010.06.010. Epub 2010 Jun 26. PMID 20579741
- [Background] Panossian A, Wikman G, Sarris J. Rosenroot (Rhodiola rosea): traditional use, chemical composition, pharmacology and clinical efficacy. Phytomedicine. 2010 Jun;17(7):481-93. doi: 10.1016/j.phymed.2010.02.002. Epub 2010 Apr 7. PMID 20378318
- [Background] Hung SK, Perry R, Ernst E. The effectiveness and efficacy of Rhodiola rosea L.: a systematic review of randomized clinical trials. Phytomedicine. 2011 Feb 15;18(4):235-44. doi: 10.1016/j.phymed.2010.08.014. Epub 2010 Oct 30. PMID 21036578
- [Background] Darbinyan V, Kteyan A, Panossian A, Gabrielian E, Wikman G, Wagner H. Rhodiola rosea in stress induced fatigue--a double blind cross-over study of a standardized extract SHR-5 with a repeated low-dose regimen on the mental performance of healthy physicians during night duty. Phytomedicine. 2000 Oct;7(5):365-71. doi: 10.1016/S0944-7113(00)80055-0. PMID 11081987
- [Background] De Bock K, Eijnde BO, Ramaekers M, Hespel P. Acute Rhodiola rosea intake can improve endurance exercise performance. Int J Sport Nutr Exerc Metab. 2004 Jun;14(3):298-307. doi: 10.1123/ijsnem.14.3.298. PMID 15256690
- [Background] Shevtsov VA, Zholus BI, Shervarly VI, Vol'skij VB, Korovin YP, Khristich MP, Roslyakova NA, Wikman G. A randomized trial of two different doses of a SHR-5 Rhodiola rosea extract versus placebo and control of capacity for mental work. Phytomedicine. 2003 Mar;10(2-3):95-105. doi: 10.1078/094471103321659780. PMID 12725561
- [Background] Spasov AA, Wikman GK, Mandrikov VB, Mironova IA, Neumoin VV. A double-blind, placebo-controlled pilot study of the stimulating and adaptogenic effect of Rhodiola rosea SHR-5 extract on the fatigue of students caused by stress during an examination period with a repeated low-dose regimen. Phytomedicine. 2000 Apr;7(2):85-9. doi: 10.1016/S0944-7113(00)80078-1. PMID 10839209
- [Background] Olsson EM, von Scheele B, Panossian AG. A randomised, double-blind, placebo-controlled, parallel-group study of the standardised extract shr-5 of the roots of Rhodiola rosea in the treatment of subjects with stress-related fatigue. Planta Med. 2009 Feb;75(2):105-12. doi: 10.1055/s-0028-1088346. Epub 2008 Nov 18. PMID 19016404
- [Background] Logan GD, Cowan WB, Davis KA. On the ability to inhibit simple and choice reaction time responses: a model and a method. J Exp Psychol Hum Percept Perform. 1984 Apr;10(2):276-91. doi: 10.1037//0096-1523.10.2.276. PMID 6232345
- [Background] Mackin RS, Horner MD. Relationship of the Wender Utah Rating Scale to objective measures of attention. Compr Psychiatry. 2005 Nov-Dec;46(6):468-71. doi: 10.1016/j.comppsych.2005.03.004. PMID 16275215